CLINICAL TRIAL: NCT03293342
Title: The Effect of a Dentist Administered Cognitive Behavioural Therapy (D-CBT) in Adult Patients With Dental Fear
Brief Title: Cognitive Behavioural Therapy and Dental Fear
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Oslo (Other)
Responsible Party: Principal Investigator, Tiril Willumsen, Professor, University of Oslo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC-2017/97
Record Dates: First submitted 2017-09-14; First posted 2017-09-26 (Actual); Last update posted 2020-11-03 (Actual); Status verified 2020-11

CONDITIONS: Dental Fear

STUDY DESIGN:
Intervention Model Description: Randomized Clinical Trial
Who Masked: Outcomes Assessor
Masking Description: Each patient receives a project number. A codebook between project number and journal number is stored at Tannhelsetjenestens kompetansesenter sør in Arendal. All data will be registered online using Nettskjema to collect data directly into Services for sensitive data (TSD). The research data from each patient will only be identified by the project number.
  All data will be stored and analysed using the TSD platform. TSD complies with the directive of privacy and electronic communication in Norway. TSD is developed and operated by USIT, the UiO centre for IT.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- D CBT (Experimental): Dentist administered cognitive behaviioral treatment
  Interventions: Behavioral: D CBT
- Control (Active Comparator): Treatment as usual
  Interventions: Combination Product: Control

INTERVENTIONS:
Behavioral: D CBT — Intervention:
  a 3-5 session treatment of dental fear.
  * Psychoeducation about anxiety
  * Exploration of the individual anxiety
  * Exposure to the frightening stimuli (no hiding, but actively showing in detail all components of dental treatment, preferably utilizing a mirror while doing treatment).
  Arms: D CBT
Combination Product: Control — Intervention:
  Traditional treatment of dental fear common sense/ benzodiazepine
  Arms: Control

SUMMARY:
The study is an RCT study comparing a 3-5 intervention treatment with dentist administered Cognitive Behavioural Therapy ( D-CBT) with a control treatment. The control treatment is a "treatment as usual" concept using premedication with benzodiazepines and a common sense approach.

The treatment will be performed in a regular dental office. The dentist is working as a regular dentist and is trained in the CBT Method.

DETAILED DESCRIPTION:
Brief Summary:

The study is an randomized clinical trial (RCT) comparing a 3-5 intervention treatment with dentist administered Cognitive Behavioural Therapy ( D-CBT) with a control treatment. The control treatment is a "treatment as usual" concept using premedication with benzodiazepines and a common sense approach.

The treatment will be performed in a regular dental office. The dentist is working as a regular dentist and is trained in the CBT Method.

Detailed Description:

Background Dental fear is common in adults and has a prevalence of about 10-25%. Approximately 2/3 of fearful patients manage to get through treatment, but with great discomfort. The remaining 1/3 avoid dental visits and some of them qualify for the diagnosis odontophobia (prevalence 1,4-7,1%).

Several studies demonstrate reduced oral health in people with dental fear and odontophobia compared to the general population.

Dental phobia often develops gradually and patients' dental health would often benefit from treatment of dental anxiety before the manifestations of phobia; before dental health deteriorate and avoidance of dental treatment has lasted too long.

Consequently, it would be beneficial if dental anxiety were effectively treated in a dentist general practice and thereby easily accessible. Thus there is a need for evidence based treatment methods for this context.

Psychological treatment of dental phobia is well documented in multidisciplinary treatment programmes were psychologists and dentists work together. However, there is a lack of psychologist resources and high cost of a treatment approach that requires 2 specialists. This emphasises the need for treatment programs of dental anxiety within dentist's competence. Dentists can, provided the right training, be successful in the utilisation of psychological techniques for the treatment of anxiety. Willumsen et al developed and tested dental anxiety treatment methods including the use of CBT interventions for use by dentists. This RCT study showed good results at post treatment, also in a 5 year follow up. Two CBT methods (applied relaxation and cognitive therapy) with contrasting principles (relaxation vs activation) were tested against nitrous oxide sedation. All three treatment approaches showed adequate effect but CBT interventions were superior in a longer time perspective. However, the treatment methods were resource demanding; requiring 10 sessions of treatment. It would therefore be beneficial to develop a shorter method of treatment that could be used by a dentist in a general practice and also to test its use within the context of a regular dental practice.

Premedication with benzodiazepines and a common sense approach including tell-show-do is the recommended and most frequent used alternative in Norway when treating this group of patients in general dental practice; Therefore the study is designed to compare the psychological intervention with these treatment modalities to explore differences in effect.

The hypothesis is that a treatment programme with D-CBT have more reduction of dental fear than traditional treatment with common sense/ premedication

The aims:

1. Test D-CBT against a combined pharmacological common sense approach in a RCT study performed in a general dental practice.
2. To explore whether demographical data, levels of dental fear, comorbidity, coping strategies or dentist-patient relation can predict treatment outcome of D-CBT.
3. To do a 1-year- and 3 year follow-up on the RCT-patients with assessment of levels of dental fear in the patient, quality of life, oral quality of life and ability to receive dental treatment.

   Methods Design The study is a randomized controlled trial. Population Patients will be recruited through written and oral information to local dentists and physicians, advertising in local newspapers or referred from a waiting list at a local dental fear clinic .

   Criteria for inclusion
   * Strong dental anxiety that affects the patients self-perceived ability to go through dental treatment
   * Age over 18
   * Agreement to all the practical arrangements of the study Criteria for exclusion
   * Substance abuse
   * Not being able to communicate fluently in Norwegian Sample size Sample size was estimated with power (1-Betta) 0,8 og type error (alfa) 5%. From these criteria sample size was calculated to 30 in each group. Drop out is expected to be about 15% giving 35 participants in each group and a total of 70 participants in the RCT-study.

   Location and operator The study will be performed in a general dental practice in Mandal, a small town in the south of Norway. All patients will be treated by the same dentist, an experienced private practitioner with an interest in treating dentally anxious patients; MSH.

   Research psychologists and dentists experienced in treating patients with dental fear have developed the dentist-based cognitive behaviour treatment method (D-CBT). D-CBT is based on existing literature.

   In addition an expert group consisting of clinical psychologists and dentists, all of which are experienced in treating dental anxiety, have assessed the practical aspects of implementing the method and manual.

   A manual describes the intervention in detail. The method will be tested in 5 patients in a pilot study.

   Randomisation procedure Patients are randomized in two groups by simple randomisation. Lists will be constructed by statistical software and treatments will then be allocated to patients in sequence using numbered opaque envelopes containing treatment allocations.

   The intervention group All patients in the D-CBT group will go through 3- 5 consultations with a duration of 60 minutes or 3 sessions of 90 minutes aimed at treating their dental anxiety. The appointments will be spaced with a maximum of 2 weeks to minimize the setback that will often occur between appointments (detailed description in appendix).

   All sessions will be videotaped throughout the study. The control group The non-intervention group will be offered premedication with midazolam during dental treatment per standard procedures. Common sense principles as communication skills, control and tell-show-do will be implemented.

   Similarities between the control and the intervention groups:
   * Building a good relation with the patient
   * Stop signal will be utilized
   * Explain and show what the dentist wants to do before doing treatment (tell-show-do)
   * The treatment should be as painless as possible

   Differences between the control and the intervention groups:

   Midazolam/tell-show-do
   * Sedation is an alternative
   * Minimalizing exposure to the patient (for example hiding instead of showing the syringe while putting the anaesthetics).

   Psycological intervention -characteristics
   * Psychoeducation about anxiety
   * Exploration of the individual anxiety
   * Exposure to the frightening stimuli (no hiding, but actively showing in detail all components of dental treatment, preferably utilizing a mirror while doing treatment).

   Data Each patient receives a project number. A codebook between project number and journal number is stored at the Specialist Center of Public Dental Health in South Norway All data will be registered online using Nettskjema to collect data directly into Services for sensitive data (TSD). The research data from each patient will only be identified by the project number.

   All data will be stored and analysed using the TSD platform. TSD complies with the directive of privacy and electronic communication in Norway. TSD is developed and operated by the University of Oslos' centre for IT (USIT).

   Only MSH and the supervisors will be given access to the data in TSD. All video recordings will be stored on encrypted memory sticks locked in a filing cabinet. The key to the filing cabinet is kept in a key cabinet locked by a code. The code is known only by the dentist (MSH) and the dental secretary (KL). The recordings will be stored up until publication of articles and TW is responsible for deleting them.

   Statistics The current project uses a traditional experimental research design to assess the research hypothesis. In order to compare differences between the 35 participants in the two research conditions the data will be analysed with regression analysis. A 2x2 repeated measures ANOVA will be used to test if the experimental condition of five sessions of D-CBT treatment is superior to the control condition of premedication and gradual habituation. A factor analytic approach will be used to assess the level of influence on the results by factors like: age; gender; social economic status and substance abuse. The statistical analysis will be completed using the IBM SPSS statistical software version 16.0.

   Measure of treatment quality and adherence All sessions will be videotaped throughout the study. At least 20% of the tapes will be viewed by the supervisors to ensure continued treatment quality and adherence to manuals.

   Measures

   Demographics data:

   The following demographics will be registered: Sex, age, Norwegian skills, civil status, children, education, work status, self-assessment of health, self-assessment of oral health and substance abuse. The patients register time since last regular appointment with a dentist.

   Level of dental anxiety: Modified Dental Anxiety Scale (MDAS) and Index of dental anxiety and fear (IDAF-4C+). .

   Measures to identify factors that may influence treatment outcome:

   Post-traumatic stress disorder: Post-traumatic stress disorder-checklist (PCL).

   Depression and anxiety: The hospital anxiety and depression scale (HADS)

   Satisfaction with life:

   The Satisfaction With Life Scale (SWLS) Oral quality of life: Oral impact on daily performance (OIDP). Patient-dentist relation: Working Alliance Inventory -12 (WAI-12).

   Coping strategies: The dental coping strategy questionnaire (DCSQ). Patient assessment of the treatment: An questionnaire containing a likert scale assessing how the patients evaluate different elements of the treatment they have received has been developed based on similar scales in comparable studies Personality traits: The Big Five Inventory

   Dental reports:

   Oral examination and assessment of x-rays. Three. dentists separately record oral health and treatment needs based on the radiographs (BWs and OPG). With access to the initial clinical recordings, the diagnostic registrations will then be discussed among the three dentists until a consensus is achieved.

   Oral Health: Decayed, missed or filled teeth (DMFT).Root-filled teeth. Remnants of roots Periradicular bone lesions. Number of third molars.

   Oral treatment needs: Number of teeth with need for restorations, periodontal treatment,root fillings, bridges , dentures and extractions.

   Ethics: The study is approved by the Regional Ethics. To make sure the quality of the intervention meets adequate standards, the dentist will go through training by qualified personnel before the study is initiated and there will be a continuous surveillance by watching videotapes of the treatment to ensure that the quality will be upheld throughout the study.

   The associate supervisor of the project, psychologist Bent Storå, will be available for guidance and help when needed.

   Researchers:

   Dentist, PhD candidate Mariann Saanum Hauge (MSH), Main supervisor professor dr. odont, Tiril Willumsen (TW), Associated supervisor clinical psychologist PhD, Bent Storå(BS), Research assistant, dental secretary Kari Laudal (KL) Financial matters The study receives financial support from the Norwegian Directorate of Health through the Specialist Center of Public Dental Health in South Norway.

ELIGIBILITY:
Inclusion Criteria:

* Strong dental anxiety that affects the patients self-perceived ability to go through dental treatment
* Age over 18
* Agreement to all the practical arrangements of the study

Exclusion Criteria:

* Substance abuse
* Not being able to communicate fluently in Norwegian

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2017-09-10 (Actual); Primary Completion 2020-11-02 (Actual); Study Completion 2022-12-20 (Estimated)

PRIMARY OUTCOMES:
Level of Dental anxiety, Dental Anxiety Scale ( MDAS) | At baseline, after 3-5 weeks of treatment, after 1 year and after 5 years
  MDAS is a 5 item scale measuring dental anxiety in a range from 5-25. Outcome measure: change in MDAS

CONTACTS AND LOCATIONS:
Overall Officials: Professor Willumsen, PdD, Principal Investigator — University of Oslo
Locations (1):
- University of Oslo, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hagglin C, Hakeberg M, Ahlqwist M, Sullivan M, Berggren U. Factors associated with dental anxiety and attendance in middle-aged and elderly women. Community Dent Oral Epidemiol. 2000 Dec;28(6):451-60. doi: 10.1034/j.1600-0528.2000.028006451.x. PMID 11106018
- [Background] Hakeberg M, Berggren U, Carlsson SG, Grondahl HG. Long-term effects on dental care behavior and dental health after treatments for dental fear. Anesth Prog. 1993;40(3):72-7. PMID 7645792
- [Background] Hakeberg M, Berggren U. Changes in sick leave among Swedish dental patients after treatment for dental fear. Community Dent Health. 1993 Mar;10(1):23-9. PMID 8495390
- [Background] Schuller AA, Willumsen T, Holst D. Are there differences in oral health and oral health behavior between individuals with high and low dental fear? Community Dent Oral Epidemiol. 2003 Apr;31(2):116-21. doi: 10.1034/j.1600-0528.2003.00026.x. PMID 12641592
- [Background] Armfield JM, Heaton LJ. Management of fear and anxiety in the dental clinic: a review. Aust Dent J. 2013 Dec;58(4):390-407; quiz 531. doi: 10.1111/adj.12118. PMID 24320894
- [Background] Davies JG, Wilson KI, Clements AL. A joint approach to treating dental phobia: a re-evaluation of a collaboration between community dental services and specialist psychotherapy services ten years on. Br Dent J. 2011 Aug 26;211(4):159-62. doi: 10.1038/sj.bdj.2011.674. PMID 21869789
- [Background] Gordon D, Heimberg RG, Tellez M, Ismail AI. A critical review of approaches to the treatment of dental anxiety in adults. J Anxiety Disord. 2013 May;27(4):365-78. doi: 10.1016/j.janxdis.2013.04.002. Epub 2013 Apr 13. PMID 23746494
- [Background] Vika M, Skaret E, Raadal M, Ost LG, Kvale G. One- vs. five-session treatment of intra-oral injection phobia: a randomized clinical study. Eur J Oral Sci. 2009 Jun;117(3):279-85. doi: 10.1111/j.1600-0722.2009.00628.x. PMID 19583756
- [Background] Willumsen T, Vassend O. Effects of cognitive therapy, applied relaxation and nitrous oxide sedation. A five-year follow-up study of patients treated for dental fear. Acta Odontol Scand. 2003 Apr;61(2):93-9. doi: 10.1080/00016350310001442. PMID 12790506
- [Background] Brahm CO, Lundgren J, Carlsson SG, Nilsson P, Hultqvist J, Hagglin C. Dentists' skills with fearful patients: education and treatment. Eur J Oral Sci. 2013 Jun;121(3 Pt 2):283-91. doi: 10.1111/eos.12017. Epub 2013 Jan 19. PMID 23659263
- [Background] Strom K, Ronneberg A, Skaare AB, Espelid I, Willumsen T. Dentists' use of behavioural management techniques and their attitudes towards treating paediatric patients with dental anxiety. Eur Arch Paediatr Dent. 2015 Aug;16(4):349-55. doi: 10.1007/s40368-014-0169-1. Epub 2015 Mar 10. PMID 25753025
- [Background] Humphris GM, Morrison T, Lindsay SJ. The Modified Dental Anxiety Scale: validation and United Kingdom norms. Community Dent Health. 1995 Sep;12(3):143-50. PMID 7584581
- [Background] Armfield JM. Development and psychometric evaluation of the Index of Dental Anxiety and Fear (IDAF-4C+). Psychol Assess. 2010 Jun;22(2):279-87. doi: 10.1037/a0018678. PMID 20528055
- [Background] Blevins CA, Weathers FW, Davis MT, Witte TK, Domino JL. The Posttraumatic Stress Disorder Checklist for DSM-5 (PCL-5): Development and Initial Psychometric Evaluation. J Trauma Stress. 2015 Dec;28(6):489-98. doi: 10.1002/jts.22059. Epub 2015 Nov 25. PMID 26606250
- [Background] Zigmond AS, Snaith RP. The hospital anxiety and depression scale. Acta Psychiatr Scand. 1983 Jun;67(6):361-70. doi: 10.1111/j.1600-0447.1983.tb09716.x. PMID 6880820
- [Background] Diener E, Emmons RA, Larsen RJ, Griffin S. The Satisfaction With Life Scale. J Pers Assess. 1985 Feb;49(1):71-5. doi: 10.1207/s15327752jpa4901_13. PMID 16367493
- [Background] Astrom AN, Haugejorden O, Skaret E, Trovik TA, Klock KS. Oral Impacts on Daily Performance in Norwegian adults: validity, reliability and prevalence estimates. Eur J Oral Sci. 2005 Aug;113(4):289-96. doi: 10.1111/j.1600-0722.2005.00225.x. PMID 16048520
- [Background] Haugejorden O, Klock KS, Astrom AN, Skaret E, Trovik TA. Socio-economic inequality in the self-reported number of natural teeth among Norwegian adults--an analytical study. Community Dent Oral Epidemiol. 2008 Jun;36(3):269-78. doi: 10.1111/j.1600-0528.2007.00367.x. PMID 18474059
- [Background] Bernson JM, Elfstrom ML, Hakeberg M. Adaptive coping strategies among adults with dental fear. Further development of a new version of the Dental Coping Strategy Questionnaire. Acta Odontol Scand. 2012 Sep;70(5):414-20. doi: 10.3109/00016357.2011.634830. Epub 2011 Nov 30. PMID 22126426
- [Background] Goldberg LR. The structure of phenotypic personality traits. Am Psychol. 1993 Jan;48(1):26-34. doi: 10.1037//0003-066x.48.1.26. PMID 8427480
- [Derived] Hauge MS, Willumsen T, Stora B. Changes in symptoms of anxiety, depression, and PTSD in an RCT-study of dentist-administered treatment of dental anxiety. BMC Oral Health. 2023 Jun 22;23(1):415. doi: 10.1186/s12903-023-03061-4. PMID 37349747
- [Derived] Hauge MS, Stora B, Vassend O, Hoffart A, Willumsen T. Dentist-administered cognitive behavioural therapy versus four habits/midazolam: An RCT study of dental anxiety treatment in primary dental care. Eur J Oral Sci. 2021 Aug;129(4):e12794. doi: 10.1111/eos.12794. Epub 2021 May 7. PMID 33960536